CLINICAL TRIAL: NCT04015895
Title: iDEFCO: Implementation of a Tool to Identify Social Weaknesses in the Cancer Care Pathway
Brief Title: Implementation of a Tool to Identify Social Weaknesses in the Cancer Care Pathway
Acronym: iDEFCO
Status: Terminated | Type: Observational
Why Stopped: low inclusion rates
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 18CH176; 2018-A03310-55 (Other: ANSM)
Record Dates: First submitted 2019-06-28; First posted 2019-07-11 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: Cancer; Social fragilities; Social inequalities; DEFCO; machine learning; cancer care pathway
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with cancer: Patient with cancer will be included. They will have to answer at DEFCO tool.
  Interventions: Other: DEFCO tool

INTERVENTIONS:
Other: DEFCO tool — The Detection of social frailties and coordination of the path of patients in cancer: a new approach by an expert computer system DEFCO tool is questionnaire to identify their social vulnerabilities. A neural network instantly identifies the patient's fragility and sends the result by email to the professionals identified in the organization of each center. These professionals then relay to the social workers in order to take care of the patient's fragility.

SUMMARY:
Social inequalities in the face of cancer are significant in all countries. They are characterized by higher mortality among people may be in the lower socioeconomic category. The care pathway may also be a source of inequality or accentuate inequalities. Socially vulnerable patients must be provided with appropriate care. It is therefore necessary to identify patients with such social vulnerabilities as early as possible and to take them into account throughout the care process. To meet this need, the DEFCO project ("Detection of social frailties and coordination of the path of patients in cancer: a new approach by an expert computer system") was designed and conducted by the Centre Hygée at the Lucien Neuwirth Cancer Institute (ICLN) in 2014 and 2015, in partnership with an industrial engineering research laboratory, the DISP ("Décision & Information pour les Systèmes de Production"). Its objective was to develop a tool for systematic screening of social fragility, involving few caregivers and making it possible to identify patients most at risk of social maladjustment. The choice was made to develop a self-administered questionnaire using tablets connected to a neural network. Since its implementation, the deployment of the DEFCO project ("Detection of social frailties and coordination of the path of patients in cancer: a new approach by an expert computer system") tool at the Lucien Neuwirth Cancer Institute (ICLN) has required several training and awareness-raising activities to strengthen the motivation of the various stakeholders. These same actors have also implemented different strategies to optimize the functioning of the tool. Developed in a specialized institution, this tool must demonstrate, in this second stage of the project, it transferability and it possibilities of implementation in other structures. It is also necessary to evaluate it in terms of it is impact, particularly on the fluidity of care pathways and on the social consequences of the disease.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the implementation of the DEFCO ("Detection of social frailties and coordination of the path of patients in cancer: a new approach by an expert computer system") social fragility tracking tool over one year.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed for cancer (solid or hematological) since 15 days maximum
* Age over 18 years
* Affiliated with or entitled to a social security scheme

Exclusion Criteria:

* Refusal to participate
* Patient unable to understand the study process
* Patient with documented history of cognitive or psychiatric disorders.
* Patient under tutorship or curatorship
* Patient not understanding French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cancer will be included.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Population reach | Months: 12
  Measured by number of actors who have been used DEFCO tool.
Population reach | Months: 12
  Measured by percentage of patient population included in relation to the target population.
Population reach | Months: 12
  Measured by rate of participation: number of patients included by physicians, proportion of patient who completed the tool, proportion of patients detected as socially fragile.
Tool adaptation by professionals | Months: 12
  Measured by number of tool variation according to centers.
Change from 6 months PACIC questionnaire result at 12 months | Months: 6, 12
  Measured by comparison Patient Assessment of Chronic Illness Care Questionnaire (PACIC) by patient at 6 and 12 months after the inclusion.
  Patient Assessment of Chronic Illness Care Questionnaire (PACIC) is a questionnaire which evaluates care during chronic illnesses with minimum score at 0 (bad care assessment) and maximum score at 130 (good care assessment).
Evaluation of effectiveness in real life by PPE | Months: 12
  Measured by comparison of Picker Patient Experience Questionnaire (PPE) between patients at 12 months after the inclusion.
  Picker Patient Experience Questionnaire (PPE) is a questionnaire which measures the patient experience with minimum score at 0 (no problem with health care access) and maximum score at 100 (problem with health care access).
Change from baseline FACT-G questionnaire result at 12 months | Months: 0, 12
  Measured by comparison Functional Assessment of Cancer Therapy-General Questionnaire (FACT-G) by patient at the baseline and 12 months after.
  Functional Assessment of Cancer Therapy-General Questionnaire (FACT-G) is a questionnaire which measures the quality of life of the patient with minimum score at 0 (low quality of life) and maximum score at 108 (high quality of life).
Change from baseline HAD questionnaire result at 12 months | Months: 0, 12
  Measured evolution of Hospital Anxiety and Depression Questionnaire (HAD) at the baseline and 12 months after.
  Hospital Anxiety and Depression Questionnaire (HAD) is a questionnaire which measures evolution of patient anxiety by 2 sub-scores :
  * Anxiety sub-score: with minimum score at 0 (no anxiety) and maximum score at 21 (anxiety)
  * Depression sub-score: with minimum score at 0 (no depression) and maximum score at 21 (depression)
Evaluation of practices effectiveness by using the tool | Months: 12
  Measured by proportion of patients who used the tool compared to patients who were included.
Evaluation of effectiveness of practices by Personalized Care Project | Months: 24
  Measured by number of social components integrated into the Personalized Care Project.
Evaluation of effectiveness of practices by identification of support systems | Months: 24
  Measured of number of support systems in each center.
Evaluation of effectiveness of practices by patient's satisfaction: questionnaire | Months: 12
  Measured by satisfaction questionnaire to the patient. Satisfaction questionnaire to the patient had 6 questions with minimum score at 0 (no contented) and maximum score at 18 (contented).
Evaluation of effectiveness of practices by caregiver's satisfaction offering the tool: questionnaire | Months: 24
  Measured by satisfaction questionnaire to the caregiver. Satisfaction questionnaire to the caregiver had 7 questions with minimum score at 0 (no contented) and maximum score at 21 (contented).
Maintenance and institutionalization | Months: 24
  Number of professionals made available for DEFCO tool.
Change from baseline interview with professional at 12 months | Months: 0, 24
  Assessed by interviews with professionals who have used DEFCO tool. Interviews with professionals will be realized at the baseline and the end at the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard +33 TARDY, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (8):
- France (8):
  - Centre Jean Perrin, Clermont-Ferrand
  - CH Emile Roux, Le Puy-en-Velay
  - Hospices Civils de Lyon - Lyon Sud, Lyon
  - Hospices Civils de Lyon, Centre Hospitalier Lyon Sud - Oncologie digestive, Lyon
  - Hospices Civils de Lyon, Groupement Hospitalier Est - Gynécologie, Lyon
  - Hospices Civils de Lyon, Groupement Hospitalier Nord - Gynécologie, Lyon
  - Chu Saint-Etienne, Saint-Etienne
  - Hôpital Privé de la Loire, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No